CLINICAL TRIAL: NCT06412198
Title: A Multicenter Phase 1b/2 Study of Adagrasib, Cetuximab, and Cemiplimab for Metastatic Colorectal Cancer Harboring KRAS G12C Mutations
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1002; NCI-2024-04127 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Colorectal Cancer; KRAS G12C Mutations
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; cemiplimab; adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lead-In (Experimental): Participants enrolled in the Lead-In phase, the dose of adagrasib participants receive will depend on when the participant join this study. The first group of participants will receive the starting dose level of adagrasib. If intolerable side effects are seen, a second group of participants will be enrolled to receive a lower dose. One (1) of these 2 doses will be chosen as the recommended dose of adagrasib.
  Interventions: Drug: Cetuximab; Drug: Cemiplimab; Drug: Adagrasib
- Expansion (Experimental): Participants enrolled in the Expansion phase, participants will receive adagrasib at the recommended dose that was found in the Lead-In phase.
  Interventions: Drug: Cetuximab; Drug: Cemiplimab; Drug: Adagrasib

INTERVENTIONS:
Drug: Cetuximab — Given by IV
  Other Names: ERBITUX
Drug: Cemiplimab — Given by IV
Drug: Adagrasib — Given by PO

SUMMARY:
To learn if the drug combination of adagrasib, cetuximab, and cemiplimab can help to control metastatic CRC with KRAS G12C mutations.

DETAILED DESCRIPTION:
Primary Objective

• To determine the objective response rate of the adagrasib, cetuximab, and cemiplimab combination for treatment of advanced KRAS G12C MT CRC that has progressed on at least one line of prior systemic chemotherapy.

Secondary Objectives

* To estimate duration of response (DOR), progression free survival (PFS), and overall survival (OS) for the combination of adagrasib, cetuximab, and cemiplimab in participants with advanced KRAS G12C MT CRC that has progressed on at least one line of prior systemic chemotherapy.
* To estimate the safety and tolerability of the combination of adagrasib, cetuximab, and cemiplimab in participants with advanced KRAS G12C MT CRC that has progressed on at least one line of prior systemic chemotherapy.

Exploratory Objectives

* To assess predictive biomarkers of response and resistance to the combination of adagrasib, cetuximab, plus cemiplimab.
* To assess mechanisms of tumor cell adaptation upon treatment with the combination of adagrasib, cetuximab, plus cemiplimab.
* To determine mechanisms of acquired resistance to the combination of adagrasib, cetuximab, plus cemiplimab.
* To assess the effect of the combination of adagrasib, cetuximab plus cemiplimab on the immune tumor microenvironment.
* To generate cell lines and participant derived xenograft (PDX) models from tumor samples.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced/metastatic microsatellite stable colorectal cancer with KRASG12C mutation with 1+ prior line(s) of therapy
* Confirmed KRASG12C mutation status. If a molecular profiling report is not available, a representative paraffin-embedded tumor block or a minimum of 10 unstained slides will be requested for retrospective KRASG12C mutation testing.
* Unresectable or metastatic disease.
* Participants must have received at least one prior line of chemotherapy for metastatic disease with progression on treatment or intolerance to therapy.
* Presence of measurable disease per RECIST 1.1
* Willingness to participate in on-study related procedures, including mandatory biopsies (one baseline and one on-treatment biopsy).
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of the proposed combination in patients <18 years of age, children are excluded from this study.
* Able to take oral medications.
* Most recent prior systemic therapy (e.g., chemotherapy, immunotherapy or investigational agent) and radiation therapy discontinued at least 7 days before first dose.
* Recovery from the treatment-related adverse effects of prior therapy at the time of enrollment to ≤ Grade 1 (excluding alopecia and prior oxaliplatin-induced neuropathy).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Laboratory values within the screening period:

  * Absolute neutrophil count ≥ 1,000/mm3 (≥ 1.0 x 109/L)
  * Platelet count ≥ 100,000/mm3 (≥ 100 x 109/L)
  * Hemoglobin ≥ 9 g/dL, in the absence of transfusions for at least 2 weeks
  * Total bilirubin ≤ 1.5x upper limit of normal (ULN) (if associated with Gilbert's disease or UGT1A1*28 homozygosity, ≤ 3x ULN)
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0x ULN (if associated with liver metastases ≤5x ULN)
  * Calculated creatinine clearance (determined as per Cockcroft-Gault) ≥ 60mL/min at screening
* Completed informed consent process, including signing of IRB-approved informed consent form.
* Willing and able to comply with clinical trial instructions and requirements. Individuals lacking the ability, based on reasonable medical judgment, to understand and appreciate the nature and consequences of participation in this study will not be eligible for participation.
* Participants who are biologically capable of having children and sexually active must agree to use an acceptable method of contraception for the duration of the treatment period and for at least 6 months after the last dose of study treatment. The Investigator will counsel the patient on selection of contraception method and instruct the participant in its consistent and correct use. Examples of acceptable forms of contraception include:

  * Oral, inserted, injected or implanted hormonal methods of contraception, provided it has been used for an adequate period of time to ensure effectiveness.
  * Correctly placed copper containing intrauterine device (IUD).
  * Male condom or female condom used WITH a spermicide.
  * Male sterilization with confirmed absence of sperm in the post-vasectomy ejaculate.
  * Bilateral tubal ligation or bilateral salpingectomy.
* The Investigator will instruct the participant to call immediately if the selected birth control method is discontinued or if pregnancy is known or suspected.

  * Note: Women are considered post-menopausal and/or not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 months ago. In case of any ambiguity, the reproductive status of the woman should be confirmed by hormone level assessment.

Exclusion Criteria:

* Prior PD1 or CTLA4 inhibition therapy
* Prior KRASG12C inhibition therapy
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Active brain metastases, unless adequately treated and participant is neurologically stable (except for residual symptoms of central nervous system treatment) for at least 2 weeks prior to enrollment without corticosteroids or are on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent)
* Ongoing need for a medication with any of the following characteristics that cannot be switched to alternative treatment within 10 days prior to study entry: known risk of QTc prolongation or Torsades de Pointes; substrate of CYP3A with a narrow therapeutic index; strong inducer or inhibitor of CYP3A and/or P-gp; strong inhibitor of BCRP; strong inhibitor or inducer of CYP2C19; and proton pump inhibitors
* Major surgery within 4 weeks of the first dose of any study drug
* History of intestinal disease or major gastric surgery likely to alter absorption of study treatment (to be determined by the treating physician)
* Pregnancy. Women of child-bearing potential must have a negative serum or urine pregnancy test during screening
* Breast-feeding or planning to breast feed during the study or within 6 months after end of treatment.
* Participants with symptomatic leptomeningeal disease.
* Major surgery within 4 weeks of first dose of any study drug.
* History of intestinal disease or major gastric surgery likely to alter absorption of study treatment, to be determined by the treating physician
* Known human immunodeficiency virus (HIV) infection or acute or chronic hepatitis B (HBV) or C (HCV) infection as tested in a CLIA certified lab using a positive HIV antibody test. For Hepatitis B and C, an antigen that is drawn and positive. Note that the following are permitted:
* Participants treated for HIV with no detectable viral load on current regimen for at least 1 month prior to randomization;
* Note: Please refer to exclusion criteria regarding drug-drug interactions of concomitant anti-HIV agents, and in particular CYP3A substrates.
* Participants with prior HBV infections who are:
* considered to have past or resolved HBV infection, defined as the presence of hepatitis B core antibody [HBcAb] and absence of hepatitis B surface antigen [HBsAg]; or
* considered to be in an inactive HBV carrier state, defined as HBsAg-positive with normal ALT, and HBV DNA < 2,000 IU/mL or < 10,000 copies/mL;
* Note: For participants in an inactive HBV carrier state or with a resolved HBV infection, the risk of HBV reactivation should be considered and the need for anti-HBV prophylaxis prior to randomization should be carefully assessed in accordance with local guidelines.
* Participants treated for HCV with no detectable viral load.
* Any serious illness, uncontrolled inter-current illness, psychiatric illness, active or uncontrolled infection, or other medical history, including laboratory results, which, in the investigator's opinion, would be likely to interfere with the participant's participation in the study, or with the interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Christine Parseghian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org